CLINICAL TRIAL: NCT03658213
Title: An Open Label, Randomised, Parallel Group, Multicentre, Non-inferiority Study to Compare ZOLADEX 10.8 mg With ZOLADEX 3.6 mg in Chinese Pre-menopausal Patients With Estrogen Receptor-Positive and HER2 Negative Early Breast Cancer
Brief Title: To Compare ZOLADEX 10.8 mg With ZOLADEX 3.6mg in Chinese Pre-menopausal ER+ HER2- Early Breast Cancer.
Acronym: LARES
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: CTP of LARES has been out of the expire date, we are trying RWS pathway for the indication expend
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8666C00004
Record Dates: First submitted 2018-06-27; First posted 2018-09-05 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Goserelin acetate; Estrogen suppression; Pre-menopausal; Zoladex
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZOLADEX 10.8 mg depot group (Experimental): • ZOLADEX 10.8 mg depot group: subcutaneous depot injection once every 12 weeks
  Interventions: Drug: ZOLADEX 10.8 mg
- ZOLADEX 3.6 mg depot group (Active Comparator): • ZOLADEX 3.6 mg depot group: subcutaneous depot injection once every 4 weeks
  Interventions: Drug: ZOLADEX 3.6mg

INTERVENTIONS:
Drug: ZOLADEX 10.8 mg — 10.8 mg depot for injection (equivalent to 10.8 mg goserelin)
  Other Names: ZOLADEX® (goserelin acetate implant) 10.8 mg
  Arms: ZOLADEX 10.8 mg depot group
Drug: ZOLADEX 3.6mg — 3.6 mg depot for injection (equivalent to 3.6 mg goserelin)
  Other Names: ZOLADEX® (goserelin acetate implant) 3.6 mg
  Arms: ZOLADEX 3.6 mg depot group

SUMMARY:
This study will recruit 168 patients in approximately 20 study centres in China.

The primary objective of this study is to examine whether ZOLADEX 10.8 mg depot is non-inferior to ZOLADEX 3.6 mg depot in terms of the suppression rate of serum estradiol (E2) to the menopausal level (≤30 pg/mL) from Week 4 through Week 24.

DETAILED DESCRIPTION:
This study will recruit 168 patients in approximately 20 study centres in China.

This open label, randomised, parallel group, multicentre study in Chinese pre menopausal patients with ER+/HER2- early breast cancer will be conducted to determine whether 3 monthly ZOLADEX 10.8 mg injection is non-inferior to monthly ZOLADEX 3.6 mg injection in terms of estradiol (E2) suppression. The study will also assess the PK, pharmacodynamics (PD), safety and tolerability of two difference strengths of ZOLADEX.

Eligible patients, as judged by the Investigator after completion of the screening tests, will be registered for this study and at the same time randomised in a 1:1 ratio to receive one of the following treatments. The study treatment must start within 7 days after randomisation.

* ZOLADEX 10.8 mg depot group: subcutaneous depot injection once every 12 weeks
* ZOLADEX 3.6 mg depot group: subcutaneous depot injection once every 4 weeks

The primary objective:

- To examine whether ZOLADEX 10.8 mg depot is non-inferior to ZOLADEX 3.6 mg depot in terms of the suppression rate of serum estradiol (E2) to the menopausal level (≤30 pg/mL) from Week 4 through Week 24.

The secondary objectives:

* To evaluate the safety and tolerability profiles of ZOLADEX 10.8 mg depot and ZOLADEX 3.6 mg depot.
* To evaluate the estradiol (E2) suppression by assessment of area under the curve (AUC) of E2 serum concentration during the 24 weeks of treatment.
* To evaluate the goserelin pharmacokinetics (PK) in Chinese patients after injection of ZOLADEX 10.8 mg depot and ZOLADEX 3.6 mg depot.
* To assess the influence on menstruous condition after injection of ZOLADEX 10.8 mg depot or ZOLADEX 3.6 mg depot.
* To assess the hormonal conditions after injection of ZOLADEX 10.8 mg depot compared with ZOLADEX 3.6 mg depot.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Women aged ≥18 at screening, in pre-menopausal status defined as:

   * Menses within 1 year before enrolment and within 3 weeks before enrolment, E2 >30 pg/mL and FSH ≤40 mIU/mL.
   * Patients who received neo/adjuvant chemotherapy before randomisation should not having chemical menopause (Patients should meet: E2>30pg/mL and FSH ≤40mIU/mL) within 12 weeks after completion of the postoperative chemotherapy.
3. Histologically confirmed ER+/HER2- primary invasive operable breast cancer (ER+ defined as at least 1% of the cells examined by immunohistochemistry testing have estrogen receptors).
4. Neoadjuvant chemotherapy and adjuvant chemotherapy prior to study enrolment are acceptable. (Please refer to Guidelines such as NCCN Clinical practice guidelines in oncology-breast cancer and CSCO-BC breast cancer guidelines for standard protocols and dosages. Please make accurate records.).
5. Have had proper surgery for primary breast cancer with no known clinical residual loco regional disease.
6. World Health Organization (WHO) performance status of 0, 1, or 2.
7. Female patients of child bearing potential and their partners, who are sexually active, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for at least 3 month after last dose of Zoladex or Tamoxifen which happens later, or they must totally/truly abstain from any form of sexual intercourse.

Exclusion Criteria:

1. Any evidence of metastatic disease.
2. Have received other previous neo/adjuvant endocrine therapy for breast cancer.
3. Other malignancy within the last 3 years except adequately treated basal cell/squamous cell carcinoma of the skin or cancer of the cervix.
4. Have any unstable complication or uncontrolled infection during screening.
5. Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, extensive bilateral lung disease on High Resolution Computed Tomography scan or any psychiatric disorder that prohibits obtaining informed consent.
6. Postmenopausal woman, defined as a woman fulfilling any of the following criteria:

   * Having undergone a bilateral oophorectomy
   * Age ≥60 years
   * Age <60 years and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression and FSH and oestradiol level in the postmenopausal range (utilising ranges from the local laboratory facility)
   * If taking tamoxifen or toremifene, and age < 60 years, then FSH and plasma oestradiol level in the postmenopausal ranges (utilising ranges from the local laboratory facility)
7. Have had a bilateral oophorectomy or ovarian irradiation.
8. HER2 overexpression or gene amplification, i.e., immunohistochemistry (IHC)3+ or fluorescence in situ hybridisation (FISH)+, where appropriate
9. Screening test results of:

   * Platelets <100 × 109/L
   * Total bilirubin >1.5 × upper limit reference range (ULRR)
   * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >2.5 × ULRR
10. Any other significantly abnormal laboratory test result at screening that would place the patient at unusual risk or confound the results of the study.
11. Patients with a relevant history of any severe concomitant disease that would place the patient at unusual risk or confound the results of the study, e.g., a strong family history of osteoporosis or severe renal or hepatic impairment.
12. Patients who, for whatever reason (e.g., confusion, infirmity, alcoholism) are unlikely to comply with study requirements as judged by the Investigator(s).
13. Patients considered by the Investigator(s) to be at risk of transmitting any infection through blood or other body fluids including the agents for acquired-immune deficiency syndrome (AIDS) or other sexually transmitted disease or hepatitis.
14. History of bleeding diathesis (i.e., disseminated intravascular coagulation [DIC] or clotting factor deficiency) or long-term anti-coagulant therapy (other than anti platelet therapy and low dose warfarin).
15. History of any hypersensitivity to active or inactive excipients of LHRH agonist or tamoxifen.
16. Patients unwilling to stop taking any drug that affects sex hormonal status, or in whom it would be inappropriate to stop.
17. Participation in another clinical study with an investigational product during the last 30 days.
18. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study centre).
19. Previous enrolment or randomisation of treatment in the present study.
20. Female patients who are pregnant or breast-feeding.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-31 (Estimated); Primary Completion 2021-11-04 (Estimated); Study Completion 2021-11-04 (Estimated)

PRIMARY OUTCOMES:
Effective inhibition rate of serum estradiol(E2) | At scheduled visits from Week 4 through Week 24.
  Percentage of participants with suppressive effect of mean serum estradiol (E2) (from 4th week to 24th week) to menopausal level (≤30 pg/mL).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From screening to 4 weeks after the completion of 24 weeks treatment period.
  All AE data will be listed and the treatment-emergence status will be flagged in the listing.
Change in Alanine aminotransferase(U/L) | At scheduled visits from screening to 24th week.
  Data for Alanine aminotransferase recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Aspartate aminotransaminase(U/L) | At scheduled visits from screening to 24th week.
  Data for Aspartate aminotransaminase recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Albumin(g/L) | At scheduled visits from screening to 24th week.
  Data for Albumin recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Alkaline phosphatase(U/L) | At scheduled visits from screening to 24th week.
  Data for Alkaline phosphatase recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Calcium(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Calcium recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Creatinine(μmoI/L) | At scheduled visits from screening to 24th week.
  Data for Creatinine recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in High density lipoprotein cholesterol(mmol/L) | At scheduled visits from screening to 24th week.
  Data for High density lipoprotein cholesterol recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Inorganic phosphate(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Inorganic phosphate recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Low density lipoprotein cholesterol(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Low density lipoprotein cholesterol recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Plasma glucose(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Plasma glucose recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Potassium(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Potassium recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Lactate dehydrogenase(U/L) | At scheduled visits from screening to 24th week.
  Data for Lactate dehydrogenase recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Triglyceride(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Triglyceride recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Sodium(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Sodium recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Total bilirubin(μmol/L) | At scheduled visits from screening to 24th week.
  Data for Total bilirubin recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Total cholesterol(mmol/L) | At scheduled visits from screening to 24th week.
  Data for Total cholesterol recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Absolute neutrophil count(/L) | At scheduled visits from screening to 24th week.
  Data for Absolute neutrophil count recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Haematocrit(vol%) | At scheduled visits from screening to 24th week.
  Data for Haematocrit recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Haemoglobin(g/L) | At scheduled visits from screening to 24th week.
  Data for Haemoglobin recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Mean cell volume(fl) | At scheduled visits from screening to 24th week.
  Data for Mean cell volume recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Platelet count(/L) | At scheduled visits from screening to 24th week.
  Data for Platelet count recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in White blood cell count (total)(/L) | At scheduled visits from screening to 24th week.
  Data for White blood cell count (total) recorded in the eCRF will be listed and summarized by treatment group and visit.
Change in Systolic Blood Pressure(mmHg) | At scheduled visits from screening to 24th week.
  Actual data and changes from baseline in Systolic blood pressure will be summarized by visit using descriptive statistics.
Change in Diastolic blood pressure(mmHg) | At scheduled visits from screening to 24th week.
  Actual data and changes from baseline in Diastolic blood pressure will be summarized by visit using descriptive statistics.
Change in Heart rate(bpm) | At scheduled visits from screening to 24th week.
  Actual data and changes from baseline in Heart rate will be summarized by visit using descriptive statistics.
To evaluate the estradiol (E2) suppression by assessment of area under the curve (AUC) of E2 serum concentration. | At scheduled visits from screening to 24th week.
  Area under the curve (AUC) of E2 serum concentration during 24 weeks of treatment
Observed maximum Goserelin plasma concentration (Cmax) | At scheduled visits from treatment start to treatment completion (week 24th).
  Only for PK subgroup; derived from the individual goserelin plasma concentration-time profiles following the first dose of study drug.
Time to maximum Goserelin plasma concentration (tmax) | At scheduled visits from treatment start to treatment completion (week 24th).
  Only for PK subgroup; derived from the individual goserelin plasma concentration-time profiles following the first dose of study drug.
Area under the Goserelin plasma concentration-time curve from time zero to time of the last measurable concentration (AUCt) | At scheduled visits from treatment start to treatment completion (week 24th).
  Only for PK subgroup; derived from the individual goserelin plasma concentration-time profiles following the first dose of study drug.
Area under the Goserelin plasma concentration-time curve from time zero to 4 weeks (AUC (0-4 weeks)) | At scheduled visits from treatment start to 4 Weeks.
  Only for 3.6 mg PK subgroup; derived from the individual goserelin plasma concentration-time profiles following the first dose of study drug.
Area under the Goserelin plasma concentration-time curve from time zero to 12 weeks (AUC (0-12 weeks)) | At scheduled visits from treatment start to 12 Weeks.
  Only for 10.8 mg PK subgroup; derived from the individual goserelin plasma concentration-time profiles following the first dose of study drug.
Trough concentration (Ctrough) | At scheduled visits from treatment start to treatment completion (24th week).
  Goserelin plasma concentration of pre-dose sample during multiple dose period.
The rate of participants who had menstruation. | At scheduled visits from screening to treatment completion (24th week), approximately 27 weeks.
  The proportion of subjects who had menstruation at each time point will be summarized by treatment group.
E2 serum concentrations | At scheduled visits from screening to treatment completion (24th week), approximately 27 weeks.
  E2 concentration at each visit will be listed and summarized for each treatment group using descriptive statistics. Mean E2 concentration versus time plots and individual FSH concentration versus time plots will be presented.
FSH serum concentrations | At scheduled visits from screening to treatment completion (24th week), approximately 27 weeks.
  FSH concentration at each visit will be listed and summarized for each treatment group using descriptive statistics. Mean FSH concentration versus time plots and individual FSH concentration versus time plots will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei JIANG, Principal Investigator — 307 Hospital of PLA
Locations (9):
- China (9):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided